CLINICAL TRIAL: NCT06130215
Title: Evaluation on Glycemic Control Using Two Different Meal Announcement Plans in Adolescents With Type 1 Diabetes on Minimed 780G Hybrid Closed Loop System
Brief Title: Simple Meal Management Using Automated Insulin Delivery System
Acronym: SMMAID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidra Medicine (Other)
Responsible Party: Principal Investigator, Goran Petrovski, Senior Attending Physcian, Prof, MD, PhD, Sidra Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2035754
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Meal Management; Automated Insulin Delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fix meal annoucement with three presets of carbohydrates (Experimental): simple meal management
  Interventions: Other: Simple meal management
- Flex meal annoucement with precise carbohydrate counting (Active Comparator): precise meal management
  Interventions: Other: Precise meal management

INTERVENTIONS:
Other: Simple meal management — * Regular meal: Total Carbs per Day x 0.6 / 3
  * Large meal: Total Carbs per Day x 0.6 / 3 x 1.5
  * Small (Snack) meal: Total Carbs per Day x 0.6 / 3 x 1.5
  Arms: Fix meal annoucement with three presets of carbohydrates
Other: Precise meal management — precise carbohydrate counting for each meal
  Arms: Flex meal annoucement with precise carbohydrate counting

SUMMARY:
Carbohydrate counting is an essential component of diabetes management in both adults and children, and together with an intensive insulin plan and increased blood glucose monitoring was associated with lower HbA1c. Carbohydrate counting is perceived as one of the most burdensome tasks in T1D and is frequently done inconsistently and with poor accuracy A recent analysis confirms that MiniMed™ Advaced Hybrid closed loop (AHCL) system is designed for optimal performance with meal announcement. Nonetheless, when meals containing < 80 grams of carbohydrates are consumed with announcement of meals at will, there is a slight reduction in the number of daily boluses with no decline in glycemic control, yet markedly less diabetes related distress and improved treatment satisfaction TIR of 78.1% in unannounced meals compared with 78.8% with announced meals .

DETAILED DESCRIPTION:
We aim to compare glucose control in adolescents with Type 1 Diabetes (T1D) without carbohydrate counting skills that use simplified meal announcement to those with carbohydrate counting skills with regular meal announcement by carbohydrates, both using MiniMed 780G system.

This study is observational, two arm, single-center, clinical investigation in subjects with type 1 diabetes on AHCL insulin pump in a period of 3 months, with extension of another 9 months.

A total of 34 individuals (age 12-17 years) will be enrolled to reach 30 individuals who will complete the 3 months study.

Participants will be assigned in two groups based on score of the Carbohydrate Assessment Tool (appendix):

* Group 1(Flex), Regular Clinical Protocol, 17 participants (Score>7)
* Group 2, (Fix), Simplified Clinical Protocol, 17 participants (Score<4) If the score is between 5-6, another training session for carbohydrate counting will be offered to the participants and assessment will be performed again to assign the participant to the each group.

After reviewing the patient's eligibility and interest, the investigators will obtain informed consent and assent as appropriate and will start the clinical process for initiating an insulin pump, which is typically done with pre-pump classes. A clinically obtained HbA1c assessment will be performed via fingerstick and DCA 2000 at baseline and 3 months during the study.

Collection of demographics and medical history, data for diabetes devices (eg meters, sensors, pumps) and brief clinical physical exam including vital signs and skin assessment will be obtained via Hospital Electronic Medical File (Cerner Millennium) and will be kept as electronic data on a separate research server.

Recruitment process All patients will be recruited during the regular clinic visits at Endocrine Clinics at Sidra Medicine in Doha. The principal investigator will evaluate if the patient meets the inclusion criteria during the regular clinic visits. Patients will be chosen first-come first-served, until 34 patients are reached. A research assistant will explain the study protocol and give patient and parent information in a confidential environment, where parents and patients will have the opportunity to ask questions about the study. Obtaining the informed consent will be ensured with participant privacy, giving adequate information about the study in a language understandable for potential subject, as well providing adequate opportunity to the subject to consider all options. The principal investigator will stress that this study is on a voluntary basis and there will be no impact on continuity of care for patients who will decide not to participate in this study. They will also be able to take the documents home, to consider their possible inclusion in the study. Parents & patients will also be able to discuss any issues or concerns or ask for clarification with the PI before including the child in the study. All subjects' questions and concerns will be answered and will be provided with necessary information. The research team will be assured of subject comprehension of the information provided.

Once the patient and parent decide to progress to inclusion within the study the research assistant will arrange a meeting for further explanation of the study protocol. Principal investigator will stress again that this study is on voluntary basis and there will be no impact on diabetes care if they decided not to participate in the study. If parents and patients have questions, those will be answered and if they need more time to decide, the research assistant will arrange another meeting. If parents and patients agree to participate in the study, consent/assent will be obtained, as required. Extra time can also be given should parents and patients decide to further consider their inclusion in the study and to sign the required consent/assent forms. Medical history, Medication history, Physical exam with Vital signs, concomitant medication will be also collected at the regular clinic visit Adverse Events in terms of hypoglycemia and hyperglycemia will be also considered on this visit and all following visits.

Base line assessment and the following variables checked at baseline:

* Age, yrs
* Gender
* Weight, kg
* Height, cm
* Duration of diabetes, yrs
* Therapy (Multiple dily injections +Self monitoring of blood glucsoe, multiple daily injections and glucose sensor, insulin pump or sensor augmented pump)
* TDD, U/(kg/d)
* HbA1c, %

Questionnaire (baseline) will be performed for both participants and parents(caregivers):

* The Diabetes Strengths and Resilience Measure for Adolescents with Type 1 Diabetes (DSTAR-Teen) (participant)
* The Brief Illness Perception Questionnaire (participant)
* PedsQL Diabetes Module Version 3.0 Child Report (participant)
* PedsQL Diabetes Module Version 3.0 Parent for Child Report (parent/caregiver)

Carbohydrate assessment tool will be given to participants (appendix) in order to evaluate the carbohydrate counting skills. This tool is already used as standard clinical practice at our department. The tool is based on 7 questions with a total score of 10. There are 3 grades:

* <4, no carbohydrate counting skills.
* 5-6, in between.
* >7, carbohydrate skills. If the score is 5 or 6, another training session will be offered to the participants in order to learn carbohydrate counting, and then the assessment will be performed again to assign the patient into the group.

Participants will be assigned in two groups based on score of the Carbohydrate Assessment Tool (appendix):

Group 1(Flex), Regular Clinical Protocol, 17 participants (Score>7) Group 2, (Fix), Simplified Clinical Protocol, 17 participants (Score<4)

Pump School: Visit 2,3 and 4 On the following visits, training on the insulin pump will be delivered to the participants.

AHCL system training. Two to four individuals and their parents/guardians will attend the group training sessions. Each session was provided by diabetes educators from 12pm to 3pm. CGM will be initiated the first day of the training, for education and observational purposes and for baseline data collection (no insulin delivery by the pump).

The program included five sessions of three hours on three consecutive days: Day 1- pump menus and icons, understanding CGM graph, education in sensor calibration and sensor insertion, MiniMed Mobile App and Carelink Connect application; Day 2- Operational modes and readiness, bolus wizard use, infusion set and reservoir change; Day 3- hypoglycemia, hyperglycemia, exercise and travel management, temporary target use; Day 4- manual Mode insulin start & final evaluation of participants' ability to handle the advanced hybrid closed loop (HCL) system.

Day 5 - Smartguard start review of manual mode report, changes to pump settings as required smartguard exits and troubleshooting.

Timing of the long-acting insulin injection will be moved two hours ahead each day during training sessions, to reach 12pm the day before the AHCL system initiation as Sensor Augmented Pump (SAP), to avoid the use of temporary basal at insulin pump initiation.

Pump school Day 4 Manual Mode Start Participants will initiate the use of the advanced HCL system in Manual Mode with suspend before low feature for 72 hours to allow the algorithm to collect insulin utilization and CGM data to establish personalized Smart Guard Auto Mode initiation parameters. Sidra's validated protocol for SAP initiation, with review of one-week CGM data will be used: in short, the protocol inputs the current insulin program (MDI), calculates a 10 to 20% reduction of total daily dose, with a 40/60 basal/bolus distribution in four or five basal rates. Insulin to carbohydrate ratio (ICR) settings utilizes the formula of 300-450/Total Daily dose (TDD) and, the formula of 90-110/TDD (mmol/l) with two Correction Factors (CF) settings, the nighttime CF set 10-20% higher than the daytime CF. Active insulin Time (AIT) is set on 3 hours, suspend before low feature is turned on with a threshold of 3.0-3.8 mmol/l (55-70 mg/dl) and glucose target range from 5.0 mmol/l to 7.2 mmol/l (90-130 mg/dl),).

Participants in both groups will initiate the SAP according to above protocol with finetuning of ICR, Basal Rates, AIT and insulin to sensitifivty factor (ISF), reviewing 7 Days of MDI+CGM data, based on clinical experience.

Pump School Day Visit 5 - Smartguard Start

AHCL Initiation and Follow up. AHCL system will be activated with the following settings:

Group 1, Precise Protocol

* Review 3 Days manual mode SAP Data
* Fine- tune ICR
* Target 100 or 110 mg/dl
* AIT: 2-3 hour
* The parameters will be set using clinical assessment and fine-tuned if needed on Follow-up visits.
* Follow up visits will be scheduled Day 7, 14,28, 56, 84 (3 months), 6, 9, & 12 Months after enabling SmartGuard (AHCL use).

Group 2, Simplified Protocol.

* Review 3 Days manual mode SAP Data
* Carb Ratio by formula 360 / TDD

  * ICR 8-10 (TDD 40-60)
  * ICR 5-7 (TDD >60)
* Target 100 mg/dl
* AIT: 2 hours
* The parameters will be fixed and fine-tuned only in case of hypoglycemia on Follow-up visits.
* Follow up visits will be scheduled on Day 7, 14, 28, 56 and In clinic Visit on Day 84 (3 months), 6, 9,& 12 Months after enabling SmartGuard (AHCL use).
* Meals: Thee sets of meal set of meals announcement carbs will be provided. Calculation will be provided by the following formula:

  * Regular meal: Total Carbs per Day x 0.6 / 3
  * Large meal: Total Carbs per Day x 0.6 / 3 x 1.5
  * Small (Snack) meal: Total Carbs per Day x 0.6 / 3 x 1.5 Total carbs per day will be calculated as average on 7-days Food Logbook diary, provided by participant, during the 7-day run in period.

No restriction in dietary intake or daily activities will be advised during the study. Clinical and technical support will be available at all times with text messaging and phone calls during the study. Standard local hypoglycemia and hyperglycemia treatment guidelines will be followed.

Smartguard Review at Day 7 & Day 14 The patient/family will upload data into the CareLink system, and the data will be reviewed by a member of the clinical team. Adjustments to system settings will be suggested to the family as clinically appropriate (system settings in Group 1, based on clinical judgement, and system settings in Group 2, only in case of hypoglycemia). The rationale for system setting adjustments will be documented.

Smartguard Review at Day 28, 56 & 84 The patient/family will upload data into the CareLink system, and the data will be reviewed by a member of the clinical team. Adjustments to system settings will be suggested to the family as clinically appropriate (system settings in Group 1, based on clinical judgement, and system settings in Group 2, only in case of hypoglycemia). The rationale for system setting adjustments will be documented.

HbA1c will be measured with point of care DCA Vantage Analyzer (Siemens, Erlangen, Germany) at baseline and at the end of the study.

Questionnaires (follow up) will be performed for both participants and parents(caregivers) at day 84.

Extension phase 9 months Smartguard Review at Day 168, 252 & 336 The patient/family will upload data into the CareLink system, and the data will be reviewed by a member of the clinical team. Adjustments to system settings will be suggested to the family as clinically appropriate (system settings in Group 1, based on clinical judgement, and system settings in Group 2, only in case of hypoglycemia). The rationale for system setting adjustments will be documented.

HbA1c will be measured with point of care DCA Vantage Analyzer (Siemens, Erlangen, Germany) at each visit.

Questionnaires (follow up) will be performed for both participants and parents(caregivers) at the end of the study (Day 336) from the initiation of AHCL system.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes >1 year prior to consent date. Diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
2. Age 12 and above at the initiation of the system
3. Total daily insulin use of great than 8.0 units per day over a 1-week period
4. Willing and able (access to internet from home) to download information into the Medtronic CareLink software
5. Clinically able to start the AHCL system

Exclusion Criteria:

1. Pregnancy
2. Untreated diabetes retinopathy, or other causes that in the investigator's opinion , precludes the individual from participating in the trial.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Hba1c | 3 months
  Change in %
Time in Range (70-180mg/dl) | 3 months
  Change in %
Time below Range (<54mg/dl and <70mg/dl) | 3 months
  Change in %
Time above Range (>180mg/dl and >250mg/dl) | 3 months
  Change in %

SECONDARY OUTCOMES:
Total Daily insulin dose | 3 months
  Change in units per day
Autocorrection insulin dose | 3 months
  Change in units per day
Severe hypoglycemia | 3 months
  number of events during the 3 months
Diabetic Ketoacidosis | 3 months
  number of events during the 3 months

OTHER OUTCOMES:
Ped Quality of Life Survey | 3 months
  Total score

CONTACTS AND LOCATIONS:
Overall Officials: Goran Petrovski, PhD, Principal Investigator — Sidra Medicine
Locations (1):
- Sidra Medicine, Doha, Qa, Qatar

IPD SHARING:
Plan to Share IPD: No
Institution policy

REFERENCES:
- [Background] Bosi E, Choudhary P, de Valk HW, Lablanche S, Castaneda J, de Portu S, Da Silva J, Re R, Vorrink-de Groot L, Shin J, Kaufman FR, Cohen O; SMILE Study Group. Efficacy and safety of suspend-before-low insulin pump technology in hypoglycaemia-prone adults with type 1 diabetes (SMILE): an open-label randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Jun;7(6):462-472. doi: 10.1016/S2213-8587(19)30150-0. Epub 2019 Apr 29. PMID 31047902
- [Background] Nathanson D, Svensson AM, Miftaraj M, Franzen S, Bolinder J, Eeg-Olofsson K. Effect of flash glucose monitoring in adults with type 1 diabetes: a nationwide, longitudinal observational study of 14,372 flash users compared with 7691 glucose sensor naive controls. Diabetologia. 2021 Jul;64(7):1595-1603. doi: 10.1007/s00125-021-05437-z. Epub 2021 Mar 27. PMID 33774713
- [Background] Tornese G, Carletti C, Giangreco M, Nistico D, Faleschini E, Barbi E. Carbohydrate Tolerance Threshold for Unannounced Snacks in Children and Adolescents With Type 1 Diabetes Using an Advanced Hybrid Closed-Loop System. Diabetes Care. 2022 Jun 2;45(6):1486-1488. doi: 10.2337/dc21-2643. PMID 35522033
- [Background] Arrieta A, Battelino T, Scaramuzza AE, Da Silva J, Castaneda J, Cordero TL, Shin J, Cohen O. Comparison of MiniMed 780G system performance in users aged younger and older than 15 years: Evidence from 12 870 real-world users. Diabetes Obes Metab. 2022 Jul;24(7):1370-1379. doi: 10.1111/dom.14714. Epub 2022 May 12. PMID 35403792
- [Background] Silva JD, Lepore G, Battelino T, Arrieta A, Castaneda J, Grossman B, Shin J, Cohen O. Real-World Performance of the MiniMed 780G System: First Report of Outcomes from 4120 Users. Diabetes Technol Ther. 2022 Feb;24(2):113-119. doi: 10.1089/dia.2021.0203. PMID 34524003
- [Background] Bell KJ, Barclay AW, Petocz P, Colagiuri S, Brand-Miller JC. Efficacy of carbohydrate counting in type 1 diabetes: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2014 Feb;2(2):133-40. doi: 10.1016/S2213-8587(13)70144-X. Epub 2013 Oct 25. PMID 24622717
- [Background] Mehta SN, Quinn N, Volkening LK, Laffel LM. Impact of carbohydrate counting on glycemic control in children with type 1 diabetes. Diabetes Care. 2009 Jun;32(6):1014-6. doi: 10.2337/dc08-2068. Epub 2009 Feb 24. PMID 19244089
- [Background] Petrovski G, Al Khalaf F, Campbell J, Fisher H, Umer F, Hussain K. 10-Day structured initiation protocol from multiple daily injection to hybrid closed-loop system in children and adolescents with type 1 diabetes. Acta Diabetol. 2020 Jun;57(6):681-687. doi: 10.1007/s00592-019-01472-w. Epub 2020 Jan 17. PMID 31953687
- [Background] Petrovski G, Campbell J, Pasha M, Day E, Hussain K, Khalifa A, van den Heuvel T. Simplified Meal Announcement Versus Precise Carbohydrate Counting in Adolescents With Type 1 Diabetes Using the MiniMed 780G Advanced Hybrid Closed Loop System: A Randomized Controlled Trial Comparing Glucose Control. Diabetes Care. 2023 Mar 1;46(3):544-550. doi: 10.2337/dc22-1692. PMID 36598841